CLINICAL TRIAL: NCT01521897
Title: Prevenar Special Use-result Surveillance (Multi-center, Prospective Observational Safety Surveillance For Prevenar In Japan)
Brief Title: Prevenar Special Use-result Surveillance in Japan (Regulatory PostMarketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-4447; B1841005 (Other: Alias Study Number)
Record Dates: First submitted 2011-09-14; First posted 2012-01-31 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Pneumococcal Vaccine; Streptococcus Pneumoniae
Keywords: Pneumococcal Vaccine; Prevenar; 7-valent; Special Use-result surveillance
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 7-valent vaccine injection: Infants starting to receive Prevenar at the age of more than 2 and less than 7 months
  Interventions: Biological: 7-valent vaccine injection

INTERVENTIONS:
Biological: 7-valent vaccine injection — For primary immunization, three doses of Prevenar 0.5 mL should be injected subcutaneously with an interval of at least 27 days between each dose. For booster immunization, one dose of Prevenar 0.5 mL should be injected subcutaneously, at least 60 days after the 3rd dose.
  Other Names: Prevenar, 7vPnC

SUMMARY:
This surveillance aims to figure out 1) use-results, 2) occurrence of adverse events, and 3) factors affecting safety in terms of the safety in infants starting to receive Prevenar at the age of more than 2 and less than 7 months in routine medical practice.

This surveillance will specifically focus on the occurrence of the following:

1. Local reactions at the injection site
2. Systemic reactions for each concomitant vaccine (especially fever more than 39C°)

DETAILED DESCRIPTION:
This surveillance will be conducted using a continuous surveillance system, in which each physician enrolls patients who meet the enrollment criteria continuously until the contract sample size is reached.

ELIGIBILITY:
Inclusion Criteria:

* Infants at the age of more than 2 and less than 7 months
* Infants who have been vaccinated with Prevenar for the first time
* Infants expected to complete four vaccinations with Prevenar

Exclusion Criteria:

Vaccination with Prevenar must not be given to any of the following;

* History of evident anaphylactic reaction to any component of Prevenar or diphtheria toxoid
* Evident pyrexia
* Evident serious acute disease
* Any other infants or children ineligible for vaccination

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants starting to receive Prevenar at the age of more than 2 and less than 7 months
Sampling Method: Probability Sample
Enrollment: 1143 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Yokoyama Children's Clinic, Kasuga, Fukuoka, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X1-4447&StudyName=Prevenar%20Special%20Use-result%20Surveillance%20in%20Japan%20%28Regulatory%20PostMarketing%20Commitment%20Plan%29%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevenar™ (7-valent): Participants were vaccinated with Prevenar™ (7-valent) as follows: for primary immunization, three doses of Prevenar™ (7-valent) 0.5 mL were injected subcutaneously with an interval of at least 27 days between each dose. For booster immunization, one dose of Prevenar™ (7-valent) 0.5 mL was injected subcutaneously, at least 60 days after the third dose.
Period: Overall Study
Arm/Group | Prevenar™ (7-valent)
Started | 1143
Completed | 1120
Not Completed | 23
Not completed — Protocol Violation | 18
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: In total, 1143 participants were enrolled in this study. Of the 1143 participants, 23 participants were excluded from the baseline analysis for the reasons of protocol violation and lost to follow-up.
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
Age, Customized [Number; unit: Participants] — Participants were vaccinated with Prevenar™ (7-valent) according to the Japanese package insert (age in months at the first vaccination).
  Participants
    2 to 4 < Months | 528
    4 to 6 < Months | 516
    6 to 7 < Months | 76
Sex: Female, Male [Count of Participants; unit: Participants] — Participants were vaccinated with Prevenar™ (7-valent) according to the Japanese package insert.
  Participants
    Female | 550
    Male | 570

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Reactions
Description: An adverse reaction was any untoward medical occurrence which was considered to be related to Prevenar™ (7-valent) in a participant who received Prevenar™ (7-valent). Relatedness to Prevenar™ (7-valent) was assessed by the sponsor (Pfizer Japan Inc.).
Time Frame: 28 days
Population: The safety analysis population comprised of participants who had received Prevenar™ (7-valent) at least once and provided the safety data and who did not meet the exclusion criteria for the safety analysis.
Measure: Number; unit: participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
participants | 126

2. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
participants | 20

3. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions (erythema, induration, tenderness, and warmth) were defined by preferred terms of MedDRA/J version 16.0 as follows: erythema for "injection site erythema"; induration for "injection site erythema" and "injection site swelling"; tenderness for "injection site pain"; and warmth for "injection site warmth".
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
Participants
  Erythema | 46
  Induration | 59
  Tenderness | 0
  Warmth | 1

4. Secondary Outcome: Number of Participants With Systemic Reactions (Pyrexia of Over 39C°) by Pattern of Concomitant Vaccination
Description: Number of participants with pyrexia (MedDRA/J version 16.0 preferred terms) of over 39C° at each vaccination time (first to fourth) was counted by each pattern of concomitant vaccination. The concomitant vaccines (CVs) used in this survey were; vaccines against Haemophilus influenzae type b (Hib), diphtheria and tetanus toxoids and pertussis (DPT), measles and rubella (MR), influenza (Flu), bacille Calmette-Guérin (BCG), vesicular stomatitis Indiana virus (VSV), Mumps, Hepatitis B (HB); and oral polio vaccine (OPV) and inactivated polio vaccine (IPV).
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
Participants
  No CVs: 1st (n =184) | 1
  No CVs: 2nd (n =166) | 1
  No CVs: 3rd (n =203) | 1
  No CVs: 4th (n =450) | 0
  Hib: 1st (n =327) | 3
  Hib: 2nd (n =207) | 0
  Hib: 3rd (n =303) | 0
  Hib: 4th (n =39) | 0
  DPT: 1st (n =176) | 1
  DPT: 2nd (n =138) | 1
  DPT: 3rd (n =72) | 0
  DPT: 4th (n =8) | 0
  MR: 1st (n =0) | 0
  MR: 2nd (n =0) | 0
  MR: 3rd (n =1) | 0
  MR: 4th (n =179) | 0
  Flu: 1st (n =0) | 0
  Flu: 2nd (n =0) | 0
  Flu: 3rd (n =3) | 0
  Flu: 4th (n =29) | 0
  BCG: 1st (n =10) | 0
  BCG: 2nd (n =6) | 0
  BCG: 3rd (n =3) | 0
  BCG: 4th (n =0) | 0
  VSV: 1st (n =0) | 0
  VSV: 2nd (n =0) | 0
  VSV: 3rd (n =0) | 0
  VSV: 4th (n =10) | 0
  Mumps: 1st (n =0) | 0
  Mumps: 2nd (n =0) | 0
  Mumps: 3rd (n =0) | 0
  Mumps: 4th (n =3) | 0
  HB: 1st (n =0) | 0
  HB: 2nd (n =1) | 0
  HB: 3rd (n =0) | 0
  HB: 4th (n =3) | 0
  OPV: 1st (n =1) | 0
  OPV: 2nd (n =1) | 0
  OPV: 3rd (n =0) | 0
  OPV: 4th (n =2) | 0
  IPV: 1st (n =0) | 0
  IPV: 2nd (n =0) | 0
  IPV: 3rd (n =0) | 0
  IPV: 4th (n =4) | 0
  DPT + Hib: 1st (n =412) | 1
  DPT + Hib: 2nd (n =556) | 1
  DPT + Hib: 3rd (n =420) | 1
  DPT + Hib: 4th (n =34) | 1
  Hib + MR: 1st (n =0) | 0
  Hib + MR: 2nd (n =1) | 0
  Hib + MR: 3rd (n =1) | 0
  Hib + MR: 4th (n =12) | 0
  Hib + Flu: 1st (n =0) | 0
  Hib + Flu: 2nd (n =2) | 0
  Hib + Flu: 3rd (n =1) | 0
  Hib + Flu: 4th (n =5) | 1
  Hib + HB: 1st (n =1) | 0
  Hib + HB: 2nd (n =1) | 0
  Hib + HB: 3rd (n =0) | 0
  Hib + HB: 4th (n =0) | 0
  BCG + Hib: 1st (n =8) | 1
  BCG + Hib: 2nd (n =2) | 0
  BCG + Hib: 3rd (n =3) | 0
  BCG + Hib: 4th (n =0) | 0
  OPV + Hib: 1st (n =1) | 0
  OPV + Hib: 2nd (n =0) | 0
  OPV + Hib: 3rd (n =4) | 0
  OPV + Hib: 4th (n =0) | 0
  DPT + MR: 1st (n =0) | 0
  DPT + MR: 2nd (n =1) | 0
  DPT + MR: 3rd (n =0) | 0
  DPT + MR: 4th (n =0) | 0
  DPT + Flu: 1st (n =0) | 0
  DPT + Flu: 2nd (n =1) | 0
  DPT + Flu: 3rd (n =0) | 0
  DPT + Flu: 4th (n =1) | 0
  DPT + VSV: 1st (n =0) | 0
  DPT + VSV: 2nd (n =0) | 0
  DPT + VSV: 3rd (n =0) | 0
  DPT + VSV: 4th (n =2) | 0
  DPT + Mumps: 1st (n =0) | 0
  DPT + Mumps: 2nd (n =0) | 0
  DPT + Mumps: 3rd (n =0) | 0
  DPT + Mumps: 4th (n =0) | 0
  MR + VSV: 1st (n =0) | 0
  MR + VSV: 2nd (n =0) | 0
  MR + VSV: 3rd (n =0) | 0
  MR + VSV: 4th (n =3) | 0
  MR + Mumps: 1st (n =0) | 0
  MR + Mumps: 2nd (n =0) | 0
  MR + Mumps: 3rd (n =0) | 0
  MR + Mumps: 4th (n =2) | 0
  MR + HB: 1st (n =0) | 0
  MR + HB: 2nd (n =0) | 0
  MR + HB: 3rd (n =0) | 0
  MR + HB: 4th (n =1) | 0
  Flu + MR: 1st (n =0) | 0
  Flu + MR: 2nd (n =0) | 0
  Flu + MR: 3rd (n =0) | 0
  Flu + MR: 4th (n =3) | 0
  Flu + Mumps: 1st (n =0) | 0
  Flu + Mumps: 2nd (n =0) | 0
  Flu + Mumps: 3rd (n =0) | 0
  Flu + Mumps: 4th (n =1) | 0
  VSV + Mumps: 1st (n =0) | 0
  VSV + Mumps: 2nd (n =0) | 0
  VSV + Mumps: 3rd (n =0) | 0
  VSV + Mumps: 4th (n =4) | 0
  MR + VSV + Mumps: 1st (n =0) | 0
  MR + VSV + Mumps: 2nd (n =0) | 0
  MR + VSV + Mumps: 3rd (n =0) | 0
  MR + VSV + Mumps: 4th (n =34) | 0
  DPT + Hib + MR: 1st (n =0) | 0
  DPT + Hib + MR: 2nd (n =0) | 0
  DPT + Hib + MR: 3rd (n =0) | 0
  DPT + Hib + MR: 4th (n =1) | 0
  Hib + MR + VSV: 1st (n =0) | 0
  Hib + MR + VSV: 2nd (n =0) | 0
  Hib + MR + VSV: 3rd (n =0) | 0
  Hib + MR + VSV: 4th (n =1) | 0
  DPT + Hib + Mumps: 1st (n =0) | 0
  DPT + Hib + Mumps: 2nd (n =0) | 0
  DPT + Hib + Mumps: 3rd (n =1) | 0
  DPT + Hib + Mumps: 4th (n =0) | 0
  DPT + Hib + HB: 1st (n =0) | 0
  DPT + Hib + HB: 2nd (n =0) | 0
  DPT + Hib + HB: 3rd (n =1) | 0
  DPT + Hib + HB: 4th (n =0) | 0
  DPT + Hib + IPV: 1st (n =0) | 0
  DPT + Hib + IPV: 2nd (n =0) | 0
  DPT + Hib + IPV: 3rd (n =1) | 0
  DPT + Hib + IPV: 4th (n =0) | 0
  VSV + Mumps + IPV: 1st (n =0) | 0
  VSV + Mumps + IPV: 2nd (n =0) | 0
  VSV + Mumps + IPV: 3rd (n =0) | 0
  VSV + Mumps + IPV: 4th (n =2) | 0
  Hib + MR + VSV + Mumps: 1st (n =0) | 0
  Hib + MR + VSV + Mumps: 2nd (n =0) | 0
  Hib + MR + VSV + Mumps: 3rd (n =0) | 0
  Hib + MR + VSV + Mumps: 4th (n =1) | 0
  Hib + MR + Mumps + IPV: 1st (n =0) | 0
  Hib + MR + Mumps + IPV: 2nd (n =0) | 0
  Hib + MR + Mumps + IPV: 3rd (n =0) | 0
  Hib + MR + Mumps + IPV: 4th (n =1) | 0
  MR + VSV + Mumps + HB: 1st (n =0) | 0
  MR + VSV + Mumps + HB: 2nd (n =0) | 0
  MR + VSV + Mumps + HB: 3rd (n =0) | 0
  MR + VSV + Mumps + HB: 4th (n =1) | 0

5. Secondary Outcome: Number of Participants With Systemic Reactions (Pyrexia) by Pattern of Concomitant Vaccination
Description: Number of participants with pyrexia (MedDRA/J version 16.0 preferred terms) at each vaccination time (first to fourth) was counted by each pattern of concomitant vaccination. The concomitant vaccines (CVs) used in this survey were; vaccines against Haemophilus influenzae type b (Hib), diphtheria and tetanus toxoids and pertussis (DPT), measles and rubella (MR), influenza (Flu), bacille Calmette-Guérin (BCG), vesicular stomatitis Indiana virus (VSV), Mumps, Hepatitis B (HB); and oral polio vaccine (OPV) and inactivated polio vaccine (IPV).
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
participants
  No CVs: 1st (n =184) | 6
  No CVs: 2nd (n =166) | 1
  No CVs: 3rd (n =203) | 3
  No CVs: 4th (n =450) | 1
  Hib: 1st (n =327) | 8
  Hib: 2nd (n =207) | 4
  Hib: 3rd (n =303) | 1
  Hib: 4th (n =39) | 0
  DPT: 1st (n =176) | 11
  DPT: 2nd (n =138) | 3
  DPT: 3rd (n =72) | 0
  DPT: 4th (n =8) | 0
  MR: 1st (n =0) | 0
  MR: 2nd (n =0) | 0
  MR: 3rd (n =1) | 0
  MR: 4th (n =179) | 2
  Flu: 1st (n =0) | 0
  Flu: 2nd (n =0) | 0
  Flu: 3rd (n =3) | 0
  Flu: 4th (n =29) | 0
  BCG: 1st (n =10) | 0
  BCG: 2nd (n =6) | 0
  BCG: 3rd (n =3) | 0
  BCG: 4th (n =0) | 0
  VSV: 1st (n =0) | 0
  VSV: 2nd (n =0) | 0
  VSV: 3rd (n =0) | 0
  VSV: 4th (n =10) | 0
  Mumps: 1st (n =0) | 0
  Mumps: 2nd (n =0) | 0
  Mumps: 3rd (n =0) | 0
  Mumps: 4th (n =3) | 0
  HB: 1st (n =0) | 0
  HB: 2nd (n =1) | 0
  HB: 3rd (n =0) | 0
  HB: 4th (n =3) | 0
  OPV: 1st (n =1) | 0
  OPV: 2nd (n =1) | 0
  OPV: 3rd (n =0) | 0
  OPV: 4th (n =2) | 0
  IPV: 1st (n =0) | 0
  IPV: 2nd (n =0) | 0
  IPV: 3rd (n =0) | 0
  IPV: 4th (n =4) | 0
  DPT + Hib: 1st (n =412) | 15
  DPT + Hib: 2nd (n =556) | 14
  DPT + Hib: 3rd (n =420) | 3
  DPT + Hib: 4th (n =34) | 1
  Hib + MR: 1st (n =0) | 0
  Hib + MR: 2nd (n =1) | 0
  Hib + MR: 3rd (n =1) | 0
  Hib + MR: 4th (n =12) | 0
  Hib + Flu: 1st (n =0) | 0
  Hib + Flu: 2nd (n =2) | 0
  Hib + Flu: 3rd (n =1) | 0
  Hib + Flu: 4th (n =5) | 1
  Hib + HB: 1st (n =1) | 0
  Hib + HB: 2nd (n =1) | 0
  Hib + HB: 3rd (n =0) | 0
  Hib + HB: 4th (n =0) | 0
  BCG + Hib: 1st (n =8) | 1
  BCG + Hib: 2nd (n =2) | 0
  BCG + Hib: 3rd (n =3) | 0
  BCG + Hib: 4th (n =0) | 0
  OPV + Hib: 1st (n =1) | 0
  OPV + Hib: 2nd (n =0) | 0
  OPV + Hib: 3rd (n =4) | 0
  OPV + Hib: 4th (n =0) | 0
  DPT + MR: 1st (n =0) | 0
  DPT + MR: 2nd (n =1) | 0
  DPT + MR: 3rd (n =0) | 0
  DPT + MR: 4th (n =0) | 0
  DPT + Flu: 1st (n =0) | 0
  DPT + Flu: 2nd (n =1) | 0
  DPT + Flu: 3rd (n =0) | 0
  DPT + Flu: 4th (n =1) | 0
  DPT + VSV: 1st (n =0) | 0
  DPT + VSV: 2nd (n =0) | 0
  DPT + VSV: 3rd (n =0) | 0
  DPT + VSV: 4th (n =2) | 0
  DPT + Mumps: 1st (n =0) | 0
  DPT + Mumps: 2nd (n =0) | 0
  DPT + Mumps: 3rd (n =0) | 0
  DPT + Mumps: 4th (n =0) | 0
  MR + VSV: 1st (n =0) | 0
  MR + VSV: 2nd (n =0) | 0
  MR + VSV: 3rd (n =0) | 0
  MR + VSV: 4th (n =3) | 0
  MR + Mumps: 1st (n =0) | 0
  MR + Mumps: 2nd (n =0) | 0
  MR + Mumps: 3rd (n =0) | 0
  MR + Mumps: 4th (n =2) | 0
  MR + HB: 1st (n =0) | 0
  MR + HB: 2nd (n =0) | 0
  MR + HB: 3rd (n =0) | 0
  MR + HB: 4th (n =1) | 0
  Flu + MR: 1st (n =0) | 0
  Flu + MR: 2nd (n =0) | 0
  Flu + MR: 3rd (n =0) | 0
  Flu + MR: 4th (n =3) | 1
  Flu + Mumps: 1st (n =0) | 0
  Flu + Mumps: 2nd (n =0) | 0
  Flu + Mumps: 3rd (n =0) | 0
  Flu + Mumps: 4th (n =1) | 0
  VSV + Mumps: 1st (n =0) | 0
  VSV + Mumps: 2nd (n =0) | 0
  VSV + Mumps: 3rd (n =0) | 0
  VSV + Mumps: 4th (n =4) | 0
  MR + VSV + Mumps: 1st (n =0) | 0
  MR + VSV + Mumps: 2nd (n =0) | 0
  MR + VSV + Mumps: 3rd (n =0) | 0
  MR + VSV + Mumps: 4th (n =34) | 1
  DPT + Hib + MR: 1st (n =0) | 0
  DPT + Hib + MR: 2nd (n =0) | 0
  DPT + Hib + MR: 3rd (n =0) | 0
  DPT + Hib + MR: 4th (n =1) | 0
  Hib + MR + VSV: 1st (n =0) | 0
  Hib + MR + VSV: 2nd (n =0) | 0
  Hib + MR + VSV: 3rd (n =0) | 0
  Hib + MR + VSV: 4th (n =1) | 0
  DPT + Hib + Mumps: 1st (n =0) | 0
  DPT + Hib + Mumps: 2nd (n =0) | 0
  DPT + Hib + Mumps: 3rd (n =1) | 0
  DPT + Hib + Mumps: 4th (n =0) | 0
  DPT + Hib + HB: 1st (n =0) | 0
  DPT + Hib + HB: 2nd (n =0) | 0
  DPT + Hib + HB: 3rd (n =1) | 0
  DPT + Hib + HB: 4th (n =0) | 0
  DPT + Hib + IPV: 1st (n =0) | 0
  DPT + Hib + IPV: 2nd (n =0) | 0
  DPT + Hib + IPV: 3rd (n =1) | 0
  DPT + Hib + IPV: 4th (n =0) | 0
  VSV + Mumps + IPV: 1st (n =0) | 0
  VSV + Mumps + IPV: 2nd (n =0) | 0
  VSV + Mumps + IPV: 3rd (n =0) | 0
  VSV + Mumps + IPV: 4th (n =2) | 0
  Hib + MR + VSV + Mumps: 1st (n =0) | 0
  Hib + MR + VSV + Mumps: 2nd (n =0) | 0
  Hib + MR + VSV + Mumps: 3rd (n =0) | 0
  Hib + MR + VSV + Mumps: 4th (n =1) | 0
  Hib + MR + Mumps + IPV: 1st (n =0) | 0
  Hib + MR + Mumps + IPV: 2nd (n =0) | 0
  Hib + MR + Mumps + IPV: 3rd (n =0) | 0
  Hib + MR + Mumps + IPV: 4th (n =1) | 0
  MR + VSV + Mumps + HB: 1st (n =0) | 0
  MR + VSV + Mumps + HB: 2nd (n =0) | 0
  MR + VSV + Mumps + HB: 3rd (n =0) | 0
  MR + VSV + Mumps + HB: 4th (n =1) | 0

6. Other Pre Specified Outcome: Number of Participants by Month of Age at Each Vaccination Time
Description: Number of participants was counted by month of age at each vaccination time (first to fourth).
Time Frame: 28 days
Population: The analysis population comprised of participants who had received Prevenar™ (7-valent) at least once and provided the safety data and who did not meet the exclusion criteria for the safety analysis.
Measure: Number; unit: Participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
Participants
  2 to less than 3 months: 1st (n =1120) | 248
  2 to less than 3 months: 2nd (n =1083) | 5
  2 to less than 3 months: 3rd (n =1017) | 0
  2 to less than 3 months: 4th (n =836) | 0
  3 to less than 4 months: 1st (n =1120) | 280
  3 to less than 4 months: 2nd (n =1083) | 193
  3 to less than 4 months: 3rd (n =1017) | 7
  3 to less than 4 months: 4th (n =836) | 0
  4 to less than 5 months: 1st (n =1120) | 297
  4 to less than 5 months: 2nd (n =1083) | 235
  4 to less than 5 months: 3rd (n =1017) | 97
  4 to less than 5 months: 4th (n =836) | 0
  5 to less than 6 months: 1st (n =1120) | 219
  5 to less than 6 months: 2nd (n =1083) | 276
  5 to less than 6 months: 3rd (n =1017) | 207
  5 to less than 6 months: 4th (n =836) | 0
  6 to less than 7 months: 1st (n =1120) | 76
  6 to less than 7 months: 2nd (n =1083) | 213
  6 to less than 7 months: 3rd (n =1017) | 241
  6 to less than 7 months: 4th (n =836) | 0
  7 to less than 8 months: 1st (n =1120) | 0
  7 to less than 8 months: 2nd (n =1083) | 93
  7 to less than 8 months: 3rd (n =1017) | 229
  7 to less than 8 months: 4th (n =836) | 1
  8 to less than 9 months: 1st (n =1120) | 0
  8 to less than 9 months: 2nd (n =1083) | 20
  8 to less than 9 months: 3rd (n =1017) | 108
  8 to less than 9 months: 4th (n =836) | 1
  9 to less than 10 months: 1st (n =1120) | 0
  9 to less than 10 months: 2nd (n =1083) | 7
  9 to less than 10 months: 3rd (n =1017) | 45
  9 to less than 10 months: 4th (n =836) | 2
  10 to less than 11 months: 1st (n =1120) | 0
  10 to less than 11 months: 2nd (n =1083) | 3
  10 to less than 11 months: 3rd (n =1017) | 18
  10 to less than 11 months: 4th (n =836) | 1
  11 to less than 12 months: 1st (n =1120) | 0
  11 to less than 12 months: 2nd (n =1083) | 4
  11 to less than 12 months: 3rd (n =1017) | 11
  11 to less than 12 months: 4th (n =836) | 7
  12 to less than 16 months: 1st (n =1120) | 0
  12 to less than 16 months: 2nd (n =1083) | 2
  12 to less than 16 months: 3rd (n =1017) | 16
  12 to less than 16 months: 4th (n =836) | 650
  16 to less than 18 months: 1st (n =1120) | 0
  16 to less than 18 months: 2nd (n =1083) | 1
  16 to less than 18 months: 3rd (n =1017) | 2
  16 to less than 18 months: 4th (n =836) | 57
  18 to less than 24 months: 1st (n =1120) | 0
  18 to less than 24 months: 2nd (n =1083) | 0
  18 to less than 24 months: 3rd (n =1017) | 4
  18 to less than 24 months: 4th (n =836) | 88
  24 months and order: 1st (n =1120) | 0
  24 months and order: 2nd (n =1083) | 0
  24 months and order: 3rd (n =1017) | 1
  24 months and order: 4th (n =836) | 6
  Unknown: 1st (n =1120) | 0
  Unknown: 2nd (n =1083) | 31
  Unknown: 3rd (n =1017) | 31
  Unknown: 4th (n =836) | 23

7. Other Pre Specified Outcome: Number of Participants by Vaccination Sites at Each Vaccination Time
Description: Number of participants was counted by vaccination sites at each vaccination time (first to fourth).
Time Frame: 28 days
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
Participants
  Upper Arm: 1st (n =1120) | 1110
  Upper Arm: 2nd (n =1083) | 1074
  Upper Arm: 3rd (n =1017) | 1013
  Upper Arm: 4th (n =836) | 836
  Other: 1st (n =1120) | 10
  Other: 2nd (n =1083) | 9
  Other: 3rd (n =1017) | 4
  Other: 4th (n= 836) | 0

8. Other Pre Specified Outcome: Number of Participants by Pattern of Concomitant Vaccines
Description: Number of participants was counted by each pattern of concomitant vaccination at each vaccination time (first to fourth). The concomitant vaccines (CVs) used were; vaccines against Haemophilus influenzae type b (Hib), diphtheria and tetanus toxoids and pertussis (DPT), measles and rubella (MR), influenza (Flu), bacille Calmette-Guérin (BCG), vesicular stomatitis Indiana virus (VSV), Mumps, Hepatitis B (HB); and oral polio vaccine (OPV) and inactivated polio vaccine (IPV).
Time Frame: 28 days
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
participants
  No CVs: 1st (n =1120) | 184
  No CVs: 2nd (n =1083) | 166
  No CVs: 3rd (n =1017) | 203
  No CVs: 4th (n =836) | 450
  Hib: 1st (n =1120) | 327
  Hib: 2nd (n =1083) | 207
  Hib: 3rd (n =1017) | 303
  Hib: 4th (n =836) | 39
  DPT: 1st (n =1120) | 176
  DPT: 2nd (n =1083) | 138
  DPT: 3rd (n =1017) | 72
  DPT: 4th (n =836) | 8
  MR: 1st (n =1120) | 0
  MR: 2nd (n =1083) | 0
  MR: 3rd (n =1017) | 1
  MR: 4th (n =836) | 179
  Flu: 1st (n =1120) | 0
  Flu: 2nd (n =1083) | 0
  Flu: 3rd (n =1017) | 3
  Flu: 4th (n =836) | 29
  BCG: 1st (n =1120) | 10
  BCG: 2nd (n =1083) | 6
  BCG: 3rd (n =1017) | 3
  BCG: 4th (n =836) | 0
  VSV: 1st (n =1120) | 0
  VSV: 2nd (n =1083) | 0
  VSV: 3rd (n =1017) | 0
  VSV: 4th (n =836) | 10
  Mumps: 1st (n =1120) | 0
  Mumps: 2nd (n =1083) | 0
  Mumps: 3rd (n =1017) | 0
  Mumps: 4th (n =836) | 3
  HB: 1st (n =1120) | 0
  HB: 2nd (n =1083) | 1
  HB: 3rd (n =1017) | 0
  HB: 4th (n =836) | 3
  OPV: 1st (n =1120) | 1
  OPV: 2nd (n =1083) | 1
  OPV: 3rd (n =1017) | 0
  OPV: 4th (n =836) | 2
  IPV: 1st (n =1120) | 0
  IPV: 2nd (n =1083) | 0
  IPV: 3rd (n =1017) | 0
  IPV: 4th (n =836) | 4
  DPT + Hib: 1st (n =1120) | 412
  DPT + Hib: 2nd (n =1083) | 556
  DPT + Hib: 3rd (n =1017) | 420
  DPT + Hib: 4th (n =836) | 34
  Hib + MR: 1st (n =1120) | 0
  Hib + MR: 2nd (n =1083) | 1
  Hib + MR: 3rd (n =1017) | 1
  Hib + MR: 4th (n =836) | 12
  Hib + Flu: 1st (n =1120) | 0
  Hib + Flu: 2nd (n =1083) | 2
  Hib + Flu: 3rd (n =1017) | 1
  Hib + Flu: 4th (n =836) | 5
  Hib + HB: 1st (n =1120) | 1
  Hib + HB: 2nd (n =1083) | 1
  Hib + HB: 3rd (n =1017) | 0
  Hib + HB: 4th (n =836) | 0
  BCG + Hib: 1st (n =1120) | 8
  BCG + Hib: 2nd (n =1083) | 2
  BCG + Hib: 3rd (n =1017) | 3
  BCG + Hib: 4th (n =836) | 0
  OPV + Hib: 1st (n =1120) | 1
  OPV + Hib: 2nd (n =1083) | 0
  OPV + Hib: 3rd (n =1017) | 4
  OPV + Hib: 4th (n =836) | 0
  DPT + MR: 1st (n =1120) | 0
  DPT + MR: 2nd (n =1083) | 1
  DPT + MR: 3rd (n =1017) | 0
  DPT + MR: 4th (n =836) | 0
  DPT + Flu: 1st (n =1120) | 0
  DPT + Flu: 2nd (n =1083) | 1
  DPT + Flu: 3rd (n =1017) | 0
  DPT + Flu: 4th (n =836) | 1
  DPT + VSV: 1st (n =1120) | 0
  DPT + VSV: 2nd (n =1083) | 0
  DPT + VSV: 3rd (n =1017) | 0
  DPT + VSV: 4th (n =836) | 2
  DPT + Mumps: 1st (n =1120) | 0
  DPT + Mumps: 2nd (n =1083) | 0
  DPT + Mumps: 3rd (n =1017) | 0
  DPT + Mumps: 4th (n =836) | 0
  MR + VSV: 1st (n =1120) | 0
  MR + VSV: 2nd (n =1083) | 0
  MR + VSV: 3rd (n =1017) | 0
  MR + VSV: 4th (n =836) | 3
  MR + Mumps: 1st (n =1120) | 0
  MR + Mumps: 2nd (n =1083) | 0
  MR + Mumps: 3rd (n =1017) | 0
  MR + Mumps: 4th (n =836) | 2
  MR + HB: 1st (n =1120) | 0
  MR + HB: 2nd (n =1083) | 0
  MR + HB: 3rd (n =1017) | 0
  MR + HB: 4th (n =836) | 1
  Flu + MR: 1st (n =1120) | 0
  Flu + MR: 2nd (n =1083) | 0
  Flu + MR: 3rd (n =1017) | 0
  Flu + MR: 4th (n =836) | 3
  Flu + Mumps: 1st (n =1120) | 0
  Flu + Mumps: 2nd (n =1083) | 0
  Flu + Mumps: 3rd (n =1017) | 0
  Flu + Mumps: 4th (n =836) | 1
  VSV + Mumps: 1st (n =1120) | 0
  VSV + Mumps: 2nd (n =1083) | 0
  VSV + Mumps: 3rd (n =1017) | 0
  VSV + Mumps: 4th (n =836) | 4
  MR + VSV + Mumps: 1st (n =1120) | 0
  MR + VSV + Mumps: 2nd (n =1083) | 0
  MR + VSV + Mumps: 3rd (n =1017) | 0
  MR + VSV + Mumps: 4th (n =836) | 34
  DPT + Hib + MR: 1st (n =1120) | 0
  DPT + Hib + MR: 2nd (n =1083) | 0
  DPT + Hib + MR: 3rd (n =1017) | 0
  DPT + Hib + MR: 4th (n =836) | 1
  Hib + MR + VSV: 1st (n =1120) | 0
  Hib + MR + VSV: 2nd (n =1083) | 0
  Hib + MR + VSV: 3rd (n =1017) | 0
  Hib + MR + VSV: 4th (n =836) | 1
  DPT + Hib + Mumps: 1st (n =1120) | 0
  DPT + Hib + Mumps: 2nd (n =1083) | 0
  DPT + Hib + Mumps: 3rd (n =1017) | 1
  DPT + Hib + Mumps: 4th (n =836) | 0
  DPT + Hib + HB: 1st (n =1120) | 0
  DPT + Hib + HB: 2nd (n =1083) | 0
  DPT + Hib + HB: 3rd (n =1017) | 1
  DPT + Hib + HB: 4th (n =836) | 0
  DPT + Hib + IPV: 1st (n =1120) | 0
  DPT + Hib + IPV: 2nd (n =1083) | 0
  DPT + Hib + IPV: 3rd (n =1017) | 1
  DPT + Hib + IPV: 4th (n =836) | 0
  VSV + Mumps + IPV: 1st (n =1120) | 0
  VSV + Mumps + IPV: 2nd (n =1083) | 0
  VSV + Mumps + IPV: 3rd (n =1017) | 0
  VSV + Mumps + IPV: 4th (n =836) | 2
  Hib + MR + VSV + Mumps: 1st (n =1120) | 0
  Hib + MR + VSV + Mumps: 2nd (n =1083) | 0
  Hib + MR + VSV + Mumps: 3rd (n =1017) | 0
  Hib + MR + VSV + Mumps: 4th (n =836) | 1
  Hib + MR + Mumps + IPV: 1st (n =1120) | 0
  HIb + MR + Mumps + IPV: 2nd (n =1083) | 0
  Hib + MR + Mumps + IPV: 3rd (n =1017) | 0
  Hib + MR + Mumps + IPV: 4th (n =836) | 1
  MR + VSV + Mumps + HB: 1st (n =1120) | 0
  MR + VSV + Mumps + HB: 2nd (n =1083) | 0
  MR + VSV + Mumps + HB: 3rd (n =1017) | 0
  MR + VSV + Mumps + HB: 4th (n =836) | 1

9. Other Pre Specified Outcome: Number of Participants by Pattern of Concomitant Vaccination Sites
Description: Number of participants was counted by each pattern of concomitant vaccination sites at each vaccination time (first to fourth). Vaccination sites of each concomitant vaccines and that of Prevenar™ (7-valent) (PVN7) were defined as follows: upper arm, UA; upper buttock, UB; femour, F; and oral route, O; R, right; L, left; same, same side of the vaccination site of PVN7; and other, other side of the vaccination site of PVN7. PVN7 was vaccinated at upper arm if not stated otherwise. The 1st to 4th represents the first to fourth vaccination of PVN7, respectively.
Time Frame: 28 days
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Prevenar™ (7-valent)
Number analyzed (Participants) | 1120
participants
  No CVs: 1st (n =1120) | 184
  No CVs: 2nd (n =1083) | 166
  No CVs: 3rd (n =1017) | 203
  No CVs: 4th (n =836) | 450
  CV, same UA: 1st (n =1120) | 5
  CV, same UA: 2nd (n =1083) | 1
  CV, same UA: 3rd (n =1017) | 5
  CV, same UA: 4th (n =836) | 2
  CV, other UA: 1st (n =1120) | 508
  CV, other UA: 2nd (n =1083) | 351
  CV, other UA: 3rd (n =1017) | 375
  CV, other UA: 4th (n =836) | 270
  CV, same F: 1st (n =1120) | 0
  CV, same F: 2nd (n =1083) | 0
  CV, same F: 3rd (n =1017) | 2
  CV, same F: 4th (n =836) | 3
  CV, O: 1st (n =1120) | 1
  CV, O: 2nd (n =1083) | 1
  CV, O: 3rd (n =1017) | 0
  CV, O: 4th (n =836) | 2
  CVs, same UA X2: 1st (n =1120) | 0
  CVs, same UA X2: 2nd (n =1083) | 0
  CVs, same UA X2: 3rd (n =1017) | 1
  CVs, same UA X2: 4th (n =836) | 0
  CVs, same UA + other UA: 1st (n =1120) | 214
  CVs, same UA + other UA: 2nd (n =1083) | 301
  CVs, same UA + other UA: 3rd (n =1017) | 236
  CVs, same UA + other UA: 4th (n =836) | 39
  CVs, other UA X2: 1st (n =1120) | 181
  CVs, other UA X2: 2nd (n =1083) | 234
  CVs, other UA X2: 3rd (n =1017) | 167
  CVs, other UA X2: 4th (n =836) | 24
  CVs, other UA + same F: 1st (n =1120) | 11
  CVs, other UA + same F: 2nd (n =1083) | 12
  CVs, other UA + same F: 3rd (n =1017) | 7
  CVs, other UA + same F: 4th (n =836) | 5
  CVs, other UA + other F: 1st (n =1120) | 0
  CVs, other UA + other F: 2nd (n =1083) | 1
  CVs, other UA + other F: 3rd (n =1017) | 4
  CVs, other UA + other F: 4th (n =836) | 0
  CVs, other UA + O: 1st (n =1120) | 1
  CVs, other UA + O: 2nd (n =1083) | 0
  CVs, other UA + O: 3rd (n =1017) | 4
  CVs, other UA + O: 4th (n =836) | 0
  CVs, other UA + other UB: 1st (n =1120) | 2
  CVs, other UA + other UB: 2nd (n =1083) | 5
  CVs, other UA + other UB: 3rd (n =1017) | 3
  CVs, other UA + other UB: 4th (n =836) | 0
  CVs, other UA + same UB: 1st (n =1120) | 2
  CVs, other UA + same UB: 2nd (n =1083) | 2
  CVs, other UA + same UB: 3rd (n =1017) | 3
  CVs, other UA + same UB: 4th (n =836) | 0
  CVs, unknown X2: 1st (n =1120) | 1
  CVs, unknown X2: 2nd (n =1083) | 0
  CVs, unknown X2: 3rd (n =1017) | 0
  CVs, unknown X2: 4th (n =836) | 0
  CVs, same UA + other UA X2: 1st (n =1120) | 0
  CVs, same UA + other UA X2: 2nd (n=1083) | 0
  CVs, same UA + other UA X2: 3rd (n =1017) | 2
  CVs, same UA + other UA X2: 4th (n =836) | 36
  CVs, other UA + same UA X2: 1st (n =1120) | 0
  CVs, other UA + same UA X2: 2nd (n =1083) | 0
  CVs, other UA + same UA X2: 3rd (n =1017) | 1
  CVs, other UA + same UA X2: 4th (n =836) | 1
  CVs, other UA X2 + same F: 1st (n =1120) | 0
  CVs, other UA X2 + same F: 2nd (n =1083) | 0
  CVs, other UA X2 + same F: 3rd (n =1017) | 0
  CVs, other UA X2 + same F: 4th (n =836) | 1
  CVs, same UA X2 + other UA X2: 1st (n =1120) | 0
  CVs, same UA X2 + other UA X2: 2nd (n =1083) | 0
  CVs, same UA X2 + other UA X2: 3rd (n =1017) | 0
  CVs, same UA X2 + other UA X2: 4th (n=836) | 2
  CVs, other UA + same UA + other F X2: 1st (n=1120) | 0
  CVs, other UA + same UA + other F X2: 2nd (n=1083) | 0
  CVs, other UA + same UA + other F X2: 3rd (n=1017) | 0
  CVs, other UA + same UA + other F X2: 4th (n=836) | 1
  PVN7, R F; CVs, R UA + L UA: 1st (n =1120) | 0
  PVN7, R F; CVs, R UA + L UA: 2nd (n =1083) | 1
  PVN7, R F; CVs, R UA + L UA: 3rd (n =1017) | 3
  PVN7, R F; CVs, R UA + L UA: 4th (n =836) | 0
  PVN7, L F; CVs, L UA + R UA: 1st (n =1120) | 4
  PVN7, L F; CVs, L UA + R UA: 2nd (n =1083) | 8
  PVN7, L F; CVs, L UA + R UA: 3rd (n =1017) | 0
  PVN7, L F; CVs, L UA + R UA: 4th (n =836) | 0
  PVN7, F; CVs, same UA + other UA: 1st (n =1120) | 5
  PVN7, F; CVs, same UA + other UA: 2nd (n =1083) | 0
  PVN7, F; CVs, same UA + other UA: 3rd (n =1017) | 1
  PVN7, F; CVs, same UA + other UA: 4th (n =836) | 0
  PVN7, F; CVs, R UA + L UA: 1st (n =1120) | 1
  PVN7, F; CVs, R UA + L UA: 2nd (n =1083) | 0
  PVN7, F; CVs, R UA + L UA: 3rd (n =1017) | 0
  PVN7, F; CVs, R UA + L UA: 4th (n =836) | 0

ADVERSE EVENTS:
Time Frame: 28 days
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Prevenar™ (7-valent)
Serious Adverse Events (participants affected / at risk) | 20/1120
Other Adverse Events (participants affected / at risk) | 464/1120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevenar™ (7-valent) (N=1120)
Cellulitis orbital (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 3 (3)
Otitis media acute (Infections and infestations) | 4 (4)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 3 (3)
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 1 (1)
Kawasaki's disease (Vascular disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Injection site swelling (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevenar™ (7-valent) (N=1120)
Bronchitis (Infections and infestations) | 119 (119)
Exanthema subitum (Infections and infestations) | 25 (25)
Gastroenteritis (Infections and infestations) | 85 (85)
Hand-foot-and-mouth disease (Infections and infestations) | 23 (23)
Nasopharyngitis (Infections and infestations) | 77 (77)
Pharyngitis (Infections and infestations) | 79 (79)
Rhinitis (Infections and infestations) | 25 (25)
Conjunctivitis (Eye disorders) | 33 (33)
Asthma (Respiratory, thoracic and mediastinal disorders) | 25 (25)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 145 (145)
Constipation (Gastrointestinal disorders) | 33 (33)
Diarrhoea (Gastrointestinal disorders) | 27 (27)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 38 (38)
Eczema (Skin and subcutaneous tissue disorders) | 91 (91)
Asteatosis (Skin and subcutaneous tissue disorders) | 24 (24)
Injection site erythema (General disorders) | 48 (48)
Injection site swelling (General disorders) | 49 (49)
Pyrexia (General disorders) | 86 (86)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.